CLINICAL TRIAL: NCT06550037
Title: Optimize and Predict Antidepressant Efficacy for Patient With Major Depressive Disorders Using Multi-omics Analysis and AI-predictive Tool
Brief Title: Optimize and Predict Antidepressant Efficacy for Patient With MDD Using Multi-omics Analysis and AI-predictive Tool
Acronym: OPADE
Status: Recruiting | Type: Observational
Sponsor: Alessio Fasano (Other)
Collaborators: University of Siena (Other); Fundació Eurecat (Other); Perseus Biomics (Unknown); ARTIFICIAL INTELLIGENCE EXPERT SRL (Industry); Mama Health Technologies GmbH (Industry); Protobios OU (Unknown); Cephalgo (Industry); Biokeralty Research Institute (Industry); Sanitas University (Other); Accare (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); Istanbul Medipol University Hospital (Other); CEINGE (Unknown); Fondazione di ricerca biomedica EBRIS (Unknown)
Responsible Party: Sponsor-Investigator, Alessio Fasano, Clinical Director, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: Pro23479
Record Dates: First submitted 2024-07-24; First posted 2024-08-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorders; Microbiome; Metabolomic; Transcriptomics; Inflammation; Immune response profiling; Genetics; Artificial intelligence; Machine learning; Electroencephalography; Chatbot; Biomarkers; Personalized medicine
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Periodic collection of blood, stool and saliva samples from enrolled patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pediatric patients affected by MDD: 14-17 years (70 pediatric patients)
- Group 1 of adult patients affected by MDD: 18-30 years (100 adult patients)
- Group 2 of adult patients affected by MDD: 31-39 years (90 adult patients)
- Group 3 of adult patients affected by MDD: 40-50 years (90 adult patients)

SUMMARY:
OPADE is a non-profit, observational, multicenter, open-label study aimed at defining personalized treatment for Major Depressive Disorder (MDD). In particular, we will combine genetics, epigenetics, microbiome, immune response data together with anamnesis, questionnaires, electroencephalography (EEG) collected from subjects suffering MDD. Eventually, an Artificial Intelligence (AI)/Machine Learning (ML) predictive tool will be created to guide clinicians in improving MDD treatment and patient's stratification.

DETAILED DESCRIPTION:
Three hundred and fifty patients diagnosed with MDD will be enrolled for 24 months and divided into 4 groups according to age: 14-17 years (70 pediatric patients), 18-30 years (100 adult patients), 31-39 years (90 adult patients), 40-50 years (90 adult patients).

The study protocol includes 6 follow-up visits: T0 (enrollment), T1, T2, T3, T4, and T5. At each medical visit, psychometric questionnaires will be administered to the patients and contextual biological samples including blood, stool and saliva will be collected. The study will use a multi-omics approach including: metagenomic sequencing to characterize the microbiome composition; metabolomics to detect circulating metabolites; transcriptomics to quantify microRNAs; epigenomics to assess methylation variability between and within groups and immune assays to analyze the antibody immune response and inflammatory profiles (cytokines, interleukins and growth factors). Cortisol and lipoproteins will also be quantified. In parallel, cognitive assessment and emotional status will be recorded remotely by each patient via chatbot and wearable EEG devices, respectively. Specifically, the chatbot will collect patient's conversations and monitoring her/his feelings; the chat conversation will be than transformed in a machine-readable data. The EEG device is a mobile app that will also allows to associate brainwaves with patients' feelings.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Major Depressive Disorder as certified by a SCID 5 (Structured Clinical Interview for DSM-5) for DSM-S for adults and K-SADS-PL-DSM 5 (Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime for DSM 5) for adolescents.
* Currently experiencing a major depressive episode with a HAM-D (Hamilton Depression) score of 18 or greater, or alternatively, a MADRS (Montgomery-Asberg Depression Rating Scale) score of 18 or greater.
* About to start a new antidepressant.
* Not concurrently starting a new psychotropic medication.
* Age 14-50 years.
* Able to use mobile devices (smart phone, tablet).
* Willingness to provide written informed consent to participate.

Exclusion Criteria:

* Intellectual disability.
* Neurological disease (multiple sclerosis, severe neurocognitive disorder, epilepsy).
* Current psychotic disorder or mood disorder with psychotic features.
* Primary diagnosis of alcohol or substance use disorder (DSM-5).
* Patients who started concomitant psychotropic medications less than one week ago.
* Active, ongoing inflammatory diseases (such as rheumatoid arthritis and rheumatic polymyalgia). or severe and unstable physical illness (such as recent myocardial infarction).
* A history of hepatitis B or C, human immunodeficiency virus, or evidence of active tuberculosis infection or any active systemic infection within 2 weeks prior to the start of the study.
* Use of antibiotics or other medications that may have affected the composition of the microbiota during the 30 days prior to baseline.
* Pregnancy and lactation.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Major Depressive Disorders
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Identify neuroinflammatory indices | 2 years
  Several inflammatory markers such as G-CSF, GM-CSF, IFN-γ IL-10, IL-12p40, IL-15, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8/CXCL8, MCP-1/CCL2, TNF-α, TNFβ will be analysed.
Microbiome analysis | 2 years
  Identification of bacterial and fungal components.
Metabolomic analysis | 2 years
  The metabolomic analysis will involve three different groups of metabolites: 1) Intermediate of tryptophan metabolism (tryptophan, serotonin, 5-HIAA, quinurenin, quinurenic acid and other hormones and derivatives involved in the pathway) and others related to purines (paraxanthin/xanthin ratio); 2) L-acylcarnitines (including short chain, medium long-lasting acylcarnitine), with particular emphasis on laurylcarnitine and acetylcarnitine; 3) Phenolic (and related), such as phenolic acid, mandelic acid or methoxy-hydroxyphenyl glycol.
Analysis of lipoprotein profile | 2 years
  Different forms of lipoproteins will be evaluated: Apolipoproteins A1 and A2, HDL-apolipoproteins A1 and A2,free cholesterol HDL3, HDL3-apolipoprotein A1, HDL2-apolipoprotein A2, apolipoprotein A2, IDL, HDL-apolipoprotein A2, VLDL and its subtypes, VLDL2-triglycerides, VLDL3-triglyceridestriglycerides, VLDL2- cholesterol, VLDL3 cholesterol, VLDL4 cholesterol free of VLDL4, phospholipids VLDL2, Phospholipids VLDL3, Cholesterol LDL5, Cholesterol free LDL5, Phospholipids LDL5, LDL5-apolipoprotein B, HDL3 cholesterol, HDL4 cholesterol HDL4, HDL3 cholesterol free, free cholesterol HDL4, HDL3-phospholipids, HDL4-phospholipids, HDL3-apolipoprotein A1, HDL4-apolipoprotein A1, HDL3-apolipoprotein A2 and HDL4-apolipoprotein A2.
Identify immune-profile linked and epigenomic signatures | 2 years
  Methylome analysis on genomic DNA will be performed.
AI-powered diagnostics predictive tool (companion diagnostic-like) | 2 years
  Deploy an AI-powered predictive tool (companion diagnostic-like) in clinical practice for the prescription of anti-depressants. OPADE AI-powered predictive tool will be a class C medical device under the In vitro diagnostic classification.
Mood assessment through brain biomarker | 2 years
  Validate a patient tracking tool for mood assessment using brain biomarker.
Patient engagement digital tool | 2 years
  Validate a patient engagement digital tool that can be deployed in any patient community to enhance clinical study outcomes.
Discovery of a new set of biomarkers | 2 years
  Propose new set of biomarkers that can guide the development of new antidepressants
Investigation of the gut-brain-axis and of the biomarkers of interest in the context of mental diseases starting with MDD | 2 years
  Identify indices in MDD to improve diagnostic accuracy for primary prevention and patients' stratification.

CONTACTS AND LOCATIONS:
Locations (1):
- Università Degli Studi Di Siena, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: OPADE Official Website — https://opade-project.eu/